CLINICAL TRIAL: NCT07366437
Title: Evaluating the Implementation and Impact of an Enhanced SNAP-Ed Delivered Curriculum in Low-income Preschools
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Director, Child Health Research Center, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB STUDY00027835
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Vegetable Acceptance in Early Childhood; Vegetable Intake; Knowledge
Keywords: SNAP-Ed; Early Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rainbow Veggie Club (Experimental): The Rainbow Veggie Club arm is the name of the educational program provided by Penn State's Child Health Research Center.
  Interventions: Behavioral: Rainbow Veggie Club

INTERVENTIONS:
Behavioral: Rainbow Veggie Club — The CATCH EC curriculum is an evidence-based program designed to promote healthy eating, physical activity, and overall wellness in early childhood and school settings. A subset of lessons from this curriculum that focus on vegetables are implemented as part of the Rainbow Veggie Club, and additional enhancements were added to the standard CATCH lessons to specifically target vegetable exposure and acceptance. These enhancements include repeated exposure of vegetables, associative conditioning by serving vegetables alongside a familiar dip, behavioral reinforcement with non-food rewards, and integration of evaluation activities.

SUMMARY:
This evaluation project aims to assess the impact of the Penn State Child Health Research Center's final year of SNAP-Ed funded nutrition education program in low-income preschool classrooms in Pennsylvania. This project uses a combination of nutrition education, repeated exposure to a variety of vegetables, and associative conditioning (using dips to make vegetables more appealing) to improve children's knowledge, acceptance, and intake of vegetables.

DETAILED DESCRIPTION:
This evaluation project aims to assess the impact of the Child Health Research Center's final year of the SNAP-Ed funded nutrition education program in low-income preschool classrooms across Pennsylvania. This is the final year of SNAP-Ed funding in Pennsylvania (made possible by state carryforward funds) due to the elimination of this funding as a result of the 2025 Big Beautiful Bill.

The intervention program, known as the Rainbow Veggie Club, is designed to enhance children's vegetable knowledge, acceptance, and intake through a comprehensive approach that combines structured nutrition education lessons, repeated exposure to a variety of vegetables, and associative conditioning techniques such as offering low-fat dips to make vegetables more appealing. The program will be implemented in a subset of classrooms where teachers and staff will receive training and follow a lesson calendar for the 2025-2026 school year.

The consent process for children includes four communications sent home to parents/guardians within a two-week period, using both electronic and paper formats, a newsletter, a consent document, and a flyer with a QR code linking to a REDCap survey. Teachers can also participate in survey data collection, in which an implied consent process will be used.

The first data collection visit includes a pre-tasting activity and Veggie Meter measurements to assess skin carotenoid levels as an objective indicator of vegetable intake. Trained staff members will conduct the Veggie Meter protocol, which is expected to take approximately one hour per classroom of 18 children, and results will be recorded on a standardized roster organized by child ID. These procedures ensure consistent data collection and allow researchers to evaluate whether the combination of education, exposure, and conditioning strategies leads to measurable improvements in children's dietary behaviors.

Data from the pre-tasting data collection will inform which vegetable will be selected for an intake assessment in visit 2. During this visit, trained staff members will conduct individual hunger assessments and measure child intake of the selected vegetable by pre- and post-weighing each food sample. Children will have an 8-minute free access period to eat the vegetable served.

After baseline data is collected, classrooms will receive a series of educational lessons from our SNAP-Ed educators from the Coordinated Approach to Child Health (CATCH) Early Childhood curriculum. These lessons will be enhanced with repeated exposure of a variety of vegetables served alongside a dip, "Taster's Awards" and other non-food rewards, and other related materials and supplies to increase learning and engagement.

Outcome measurement (tasting, Veggie Meter, and intake assessment) is repeated after the educational program to evaluate change. In addition to child-level outcomes, feasibility and implementation data will be collected throughout the program to assess how practical and sustainable this intervention is in real-world preschool settings. These data include staff adherence to protocols, time required for each activity, supply needs, and teacher engagement. Collecting feasibility and implementation metrics is critical because it informs whether the Rainbow Veggie Club model can be scaled and replicated beyond the study classrooms, ensuring that future SNAP-Ed or similar programs can adopt evidence-based strategies that are both effective and operationally realistic.

ELIGIBILITY:
Inclusion Criteria:

* Child enrolled in a participating low-income preschool classroom
* Teacher employed in a participating low-income preschool classroom

Exclusion Criteria:

* Food allergies that would restrict the participation in the data collection procedures

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Vegetable Knowledge (questions developed for study) | From enrollment to the end of intervention (approximately 5 months)
  Children will be asked if they know the name of each vegetables served before intervention and after intervention.
Vegetable Acceptance (Tasting Assessment) | From enrollment to the end of intervention (approximately 5 months)
  Acceptance of vegetables served will be measured during a tasting assessment. Research personnel will record if child refuses or tastes each food provided and then will have child rank preference of each food tasted.
Vegetable Intake Assessment | From enrollment to the end of intervention (approximately 5 months)
  Children will be served 60g of a vegetable that has been pre-weighed. We will post-weigh to calculate exact intake.

SECONDARY OUTCOMES:
Feasibility of delivering this educational program | From enrollment to the end of intervention (approximately 5 months)
  We will measure feasibility of implementing this program in real-world setting via teacher questionnaire. This questionnaire will be developed in-house to include data specific to this educational program.
Implementation data | From enrollment to the end of intervention (approximately 5 months)
  We will collect data via questionnaire after each educational lesson related to engagement, modifications made, attendance, etc. These questions will be specific to the educational lessons of the program.

CONTACTS AND LOCATIONS:
Locations (1):
- The Learning Express, Altoona, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This is a small scale study that is evaluating the impacts of our outreach programming and is not generalizable.

REFERENCES:
- See also: Related Info — https://www.fns.usda.gov/obbb
- See also: Related Info — https://snaped.fns.usda.gov/
- See also: Related Info — https://catch.org/program/early-childhood/